CLINICAL TRIAL: NCT02941822
Title: A Phase IIA Prospective, Single-Centre, Open Label Clinical Trial to Evaluate the Safety, Tolerability and Pharmacodynamic Effects of Ambroxol in Patients With Parkinson Disease: Ambroxol in Disease Modification in Parkinson Disease
Brief Title: Ambroxol in Disease Modification in Parkinson Disease
Acronym: AiM-PD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cure Parkinson's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UCL 15/0118
Record Dates: First submitted 2016-09-05; First posted 2016-10-21 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Ambroxol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Each patient will self-administer the study drug, ambroxol (60 mg per tablet) at 5 intra-dose escalations (DE) over the duration of 6 months that will be taken three times a day, see below:
  1. Day 1-7, 60 mg
  2. Day 8-14, 120 mg
  3. Day 15-21, 180 mg
  4. Day 22-28, 300 mg
  5. Day 29-186, 420 mg
  Interventions: Drug: Ambroxol

INTERVENTIONS:
Drug: Ambroxol — Details outlines in the intervention description.
  Other Names: Brand name: Ambrosan

SUMMARY:
This study will evaluate the safety, tolerability and pharmacodynamics of ambroxol in participants with Parkinson Disease. Participants will administer ambroxol at five dose levels and will undergo clinical assessments, lumbar punctures, venepuncture, biomarker blood analysis and cognitive assessment throughout the course of the study.

DETAILED DESCRIPTION:
The AiM-PD study will recruit 20 patients (10 GBA-positive & 10 GBA-negative status) diagnosed with Parkinson disease (PD). Each patient will self-administer the study drug, ambroxol (60 mg per tablet) at 5 intra-dose escalations over the course of 6 months, as shown below:

1. Day 1-7: 60 mg three times a day
2. Day 8-14: 120 mg three times a day
3. Day 15-21: 180 mg three times a day
4. Day 22-28: 300 mg three times a day
5. Day 29-186: 420 mg three times a day

The study drug is licensed in the EU as an over-the-counter drug to treat respiratory conditions by reducing mucus production. Previous studies have shown that ambroxol can penetrate the brain in rodent and non-human primate models, and may have an effect in slowing PD. The results also indicate individuals who express the GBA mutation (increased risk of PD) are able to reduce the growth of cells that cause PD by stimulating an enzyme called glucocerebrosidase.

The study will collect cerebrospinal fluid, blood, and urine samples before, during and after the drug has been taken over a 6 month period. In these samples the Investigators will measure ambroxol drug levels, assess whether the glucocerebrosidase enzyme has been stimulated and the levels of other substances thought to be associated with the development of PD and confirm whether the study drug has penetrated the cerebrospinal fluid and CNS. The study will administer clinical and cognitive assessments to determine if there is any improvement in patient's PD symptoms. If the study proves ambroxol penetrates the CNS and replicates our current findings in the laboratory, the Investigators shall move on to a much larger drug trial to test whether the study drug may be able to slow the progression of PD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female;
2. Age ≥ 40 and ≤ 80 years of age;
3. Confirmed diagnosis of Parkinson disease at any time; and Hoehn and Yahr criteria, confirmed staged between I - III, inclusive;
4. Able and willing to provide informed consent prior to any study related assessments and procedures at screening visit 1;
5. Capable of complying with all study procedures, including fasting lumbar puncture;
6. Willing to provide a blood sample for screening genomic for Parkinson Disease related DNA analysis and/or consent to Investigators obtaining and using participants previous DNA results if applicable;
7. Willing and able to self-administer oral ambroxol medication, from day 1 to 186 (at 60 mg TID (day 1-7), 120 mg TID (day 8-14), 180 mg TID (day 15-21), 300 mg TID (day 22-28) and 420 mg TID (day 29-186));
8. Able to travel to the participating study site;
9. A female participant is eligible to participate if she is of:

   * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 consecutive months of spontaneous amenorrhea, at least 6 weeks post-surgical bilateral oophorectomy (with or without hysterectomy) or post tubal ligation. In questionable cases, menopausal status will be confirmed by demonstrating levels of follicle stimulating hormone (FSH) 25.8 - 134.8 IU/L and oestradiol < 201 pmol/l at entry.
   * Women of child-bearing potential must use accepted contraceptive methods (listed below), and must have a negative serum at screening visit 1 and urine pregnancy tests at subsequent visits if applicable. An additional pregnancy test will be performed, and results obtained, prior to administration of the first dose of ambroxol.

Accepted contraception methods:

• True abstinence: When this is in line with the preferred and usual lifestyle of the participant. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception).

Contraceptive Methods with a Failure Rate of < 1%:

* Oral contraceptive, either combined or progestogen alone;
* Injectable progestogen;
* Implants of levonorgestrel;
* Estrogenic vaginal ring;
* Percutaneous contraceptive patches;
* Intrauterine device (IUD) or intrauterine system (IUS) that meets the <1% failure rate as stated in the product label;

Please note:

* All male and female participants of child bearing potential must agree with their partners to use double-barrier birth control or abstinence while participating in the study and for 2 weeks following the last dose of the study drug.
* Participants may continue to take PD medications including glutamate antagonists, anticholinergics, dopamine agonists, Levodopa (L-DOPA and decarboxylase (DDC) inhibitor), Monoamine oxidase B (MAO-B) inhibitors catechol-O-methyltransferase (COMT) inhibitors, beta blockers, selective serotonin uptake inhibitors (SSRIS), tricyclic antidepressants (TCAs) and indomethacin.

Exclusion Criteria:

Participants are excluded from participating in this study if 1 or more of the following criteria are met:

1. Current treatment with anticoagulants (e.g. warfarin) that might preclude safe completion of the lumbar puncture and in the opinion of the Investigator;
2. Current use of investigational medicinal product or participation in another interventional clinical trial or who have done so within 30 days prior to the first dose in the current study;
3. Exposure to more than three investigational medicinal products within 12 months prior to the first dose in the current study;
4. Confirmed dysphagia that would preclude self-administration of ambroxol up to 7 tablets TID for the duration of day 1 to day 186);
5. Significant known lower spinal malformations or other spinal abnormalities that would preclude lumbar puncture;
6. History of known sensitivity to the study medication,ambroxol or its excipients (lactose monohydrate, granulated microcrystalline cellulose, copovidone and magnesium stearate) in the opinion of the investigator that contraindicates their participation;
7. History of known rare hereditary disorders of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption;
8. Evidence or history of hypersensitivity to lidocaine or its derivatives;
9. History of drug abuse or alcoholism in the opinion of the Investigator that would preclude participation in the study;
10. Donation of blood (one unit or 350 ml) within three months prior to receiving the first dose of the study drug;
11. Pregnant or breastfeeding;
12. All participants of child bearing potential in the opinion of the Investigator that would preclude participation in the study and who do not agree to use double-barrier birth control or abstinence while participating in the study and for two weeks following the last dose of study drug;
13. Any clinically significant or unstable medical or surgical condition that in the opinion of the PI or PI-delegated clinician may put the participant at risk when participating in the study or may influence the results of the study or affect the participant's ability to take part in the study, as determined by medical history, physical examinations, electrocardiogram (ECG), or laboratory tests. Such conditions may include:

    1. Impaired renal function
    2. Moderate/Severe hepatic impairment
    3. A major cardiovascular event (e.g. myocardial infarction, acute coronary syndrome, decompensated congestive heart failure, pulmonary embolism, coronary revascularisation that occurred within 6 months prior to the screening visit.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-12; Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Glucocerebrosidase and ambroxol levels in blood and cerebrospinal fluid | Day 1-186
  Assess ambroxol's central nervous system and cerebrospinal fluid penetration, and its binding to GCase by examining GCase activity & ambroxol levels at 5 intra-participant dose escalations from day 1 to day 186.

SECONDARY OUTCOMES:
Prevalence of treatment-related adverse events and abnormal investigation findings at each dose escalation level | Day 1-186
  Assess the safety and tolerability of the Glucocerebrosidase (GCase) modulating chaperone ambroxol in Parkinson disease patients with and without Gaucher gene (GBA) mutation at 5 intra-participant dose escalations from day 1 to 186.
  This will include:
  the number and proportion of subjects with AEs; assessment of clinical laboratory parameters; assessment of vital signs and ECG parameters.
Pharmacodynamic effects of ambroxol on glucocerebrosidase activity in blood and CSF | Day 1-186
Effect of ambroxol on blood and CSF biomarkers | Day 1-186
  Quantify the effects of ambroxol on biomarkers of Parkinson and neurodegeneration at 5 intra-participant dose escalations from day 1 to 186.

OTHER OUTCOMES:
Improvement in Montreal Cognitive Assessment (MoCA) and Unified Parkinson's Disease Rating Scale (UPDRS) scores | Day 1-186
Improvement in non-motor symptom assessment scale (NMSS) and non-motor symptom questionnaire (NMSQuest) scores. | Day 1-186

CONTACTS AND LOCATIONS:
Locations (1):
- Leonard Wolfson Experimental Neurology Centre Clinical Research Facility LWENC CRF, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
No, all subject's data will be anonymised.

REFERENCES:
- [Derived] Mullin S, Smith L, Lee K, D'Souza G, Woodgate P, Elflein J, Hallqvist J, Toffoli M, Streeter A, Hosking J, Heywood WE, Khengar R, Campbell P, Hehir J, Cable S, Mills K, Zetterberg H, Limousin P, Libri V, Foltynie T, Schapira AHV. Ambroxol for the Treatment of Patients With Parkinson Disease With and Without Glucocerebrosidase Gene Mutations: A Nonrandomized, Noncontrolled Trial. JAMA Neurol. 2020 Apr 1;77(4):427-434. doi: 10.1001/jamaneurol.2019.4611. PMID 31930374
- See also: AiM-PD Reference 4 — http://doi.org/10.1016/j.bcmd.2012.10.007
- See also: AiM-PD Reference 8 — http://doi.org/10.1016/S0140-6736(08)61522-6
- See also: AiM-PD Reference 11 — http://doi.org/10.1016/j.braindev.2012.05.008
- See also: AiM-PD Reference 13 — http://doi.org/10.1016/j.cell.2011.06.001
- See also: AiM-PD Reference 14 — http://doi.org/10.1136/jnnp-2012-302402